CLINICAL TRIAL: NCT02093377
Title: Treatment of Sleep Apnea Early After Myocardial Infarction With Adaptive Servo-Ventilation - a Randomized Controlled Trial
Brief Title: ASV for Sleep Apnea After Myocardial Infarction
Acronym: TEAM-ASV-I
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Throughout the COVID-19 pandemic no patient could be recruited. Patients refuse to visit the hospital for study visits.
Sponsor: University Hospital Regensburg (Other)
Collaborators: ResMed Foundation (Other)
Responsible Party: Principal Investigator, Michael Arzt, Principal Investigator, University Hospital Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol Version 6.0
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Acute Myocardial Infarction; Sleep Apnea
Keywords: acute myocardial infarction; sleep apnea; adaptive servo-ventilation
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): optimal medical therapy for the management of myocardial infarction according to the current guidelines of the European Society of Cardiology alone
- Adaptive servo-ventilation (Active Comparator): optimal medical therapy for the management of myocardial infarction according to the current guidelines of the European Society of Cardiology plus treatment of sleep apnea with adaptive servo-ventilation (ASV, most recent technology of AutoSetCS device, ResMed, Sydney, Australia). Dose: The optimal ASV settings will be determined during 1-2 nights monitored by polygraphy within 5 days after PCI.
  Interventions: Device: Adaptive servo-ventilation

INTERVENTIONS:
Device: Adaptive servo-ventilation — Adaptive servo-ventilation (ASV, most recent technology of AutoSetCS device, ResMed, Sydney, Australia)
  Other Names: ASV
  Arms: Adaptive servo-ventilation

SUMMARY:
The aim of this randomized controlled trial is to test the effect of 12 weeks Adaptive Servo-Ventilation (ASV) therapy (additionally to optimal medical management of myocardial infarction) on myocardial salvage (MSI=myocardial salvage/area at risk, primary endpoint).

DETAILED DESCRIPTION:
Primary Outcome Measure: myocardial salvage index, MSI

- To test the effect of 12 weeks of ASV (additionally to percutaneous coronary intervention, PCI, and optimal medical management of AMI) on myocardial salvage (myocardial salvage index, MSI, assessed by cardiovascular magnetic resonance imaging, CMR).

Secondary Outcome Measures:

- To test whether ASV therapy in patients with SA early after AMI decreases infarct size and improves left ventricular remodelling (myocardial salvage, microvascular obstruction change of infarct size, infarct size at 12 weeks, change of left ventricular ejection fraction (LVEF), left ventricular systolic volume (LVSV), left ventricular diastolic volume (LVDV) and LVEF at 12 weeks; assessed with CMR).

B-type natriuretic peptide (NT-proBNP)

* To test whether ASV therapy in patients with SA early after AMIimproves disease specific symptom burden (Seattle Angina Questionnaire)
* To test whether ASV therapy in patients with sleep apnea early after AMI suppresses sleep apnea (apneas and hypopneas/hour of sleep, mean oxygen saturation).
* To test whether ASV therapy in patients with sleep apnea early after AMI increases renal function (Glomerular Filtration Rate, calculated using the 4vMDRD formula).

ELIGIBILITY:
Inclusion Criteria:

1. age 18-80 years
2. first AMI (ST-elevation in ECG or acute occlusion of coronary artery)
3. Primary successful PCI achieved <24 h after symptom onset
4. SA with an AHI >=15 per hour recording time
5. written informed consent

Exclusion criteria:

1. previous myocardial infarction
2. previous myocardial revascularization (PCI or surgical)
3. LVEF <45% and central sleep apnea
4. indication for a surgical revascularisation
5. cardiogenic shock, mean supine blood pressure <60mmHg or NYHA class IV
6. implanted cardiac device or other contraindications for CMR
7. known allergies or other contraindication to contrast medium (e.g. GFR<30ml/min/1.73m²)
8. history of stroke
9. contraindications for positive airway pressure support (hypotension with mean supine BP <60mmHg, dehydration, inability to clear secretions, patients at risk for aspiration of gastric contents, severe bullous lung disease, history of pneumothorax and/or pneumomediastinum, a history of epistaxis, causing pulmonary aspiration of blood, cerebrospinal fluid leak or recent skull operations or injury) patients on or with indication for oxygen therapy, mechanical/non-invasive ventilation
10. patients on nocturnal positive airway pressure support
11. severe obstructive or restrictive airway disease
12. heart failure due to primary valve disease
13. patients awaiting heart transplantation
14. diurnal symptoms of OSA requiring immediate treatment
15. pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-02; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
myocardial salvage index, MSI | 12 weeks
  To test the effect of 12 weeks of ASV (additionally to percutaneous coronary intervention, PCI, and optimal medical management of AMI) on myocardial salvage (myocardial salvage index, MSI, assessed by cardiovascular magnetic resonance imaging, CMR).

SECONDARY OUTCOMES:
infarct size and left ventricular remodelling | 12 weeks
  To test whether ASV therapy in patients with SA early after AMI decreases infarct size and improves left ventricular remodelling (myocardial salvage, microvascular obstruction change of infarct size, infarct size at 12 weeks, change of left ventricular ejection fraction (LVEF), left ventricular systolic volume (LVSV), left ventricular diastolic volume (LVDV) and LVEF at 12 weeks; assessed with CMR).
B-type natriuretic peptide (NT-proBNP) | 12 weeks
  To test whether ASV therapy in patients with SA early after AMI reduces B-type natriuretic peptide (NT-proBNP).
disease specific symptom burden | 12 weeks
  To test whether ASV therapy in patients with SA early after AMIimproves disease specific symptom burden (Seattle Angina Questionnaire)
suppresses sleep apnea | 12 weeks
  To test whether ASV therapy in patients with sleep apnea early after AMI suppresses sleep apnea (apneas and hypopneas/hour of sleep, mean oxygen saturation).
renal function | 12 weeks
  increases renal function (Glomerular Filtration Rate, calculated using the 4vMDRD formula).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Arzt, MD, Principal Investigator — University Hospital Regensburg
Locations (5):
- Germany (5):
  - Universitätsklinikum Aachen, Aachen
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Unfallkrankenhaus Berlin, Berlin
  - Klinikum Oldenburg, Oldenburg
  - University Hospital Regensburg, Regensburg

REFERENCES:
- [Derived] Pec J, Baumert M, Fox H, Stadler S, Driendl S, Oldenburg O, Zeman F, Tanacli R, Kelle S, Buchner S, Arzt M. Effects of treatment with minute-ventilation triggered adaptive servo-ventilation early after acute myocardial infarction on nocturnal hypoxaemic burden: results from TEAM-ASV I. Sleep. 2026 Jan 8:zsaf411. doi: 10.1093/sleep/zsaf411. Online ahead of print. PMID 41504368
- [Derived] Pec J, Fox H, Stadler S, Hetzenecker A, Oldenburg O, Koller M, Zeman F, Buchner S, Wagner S, Arzt M; TEAM-ASV I Investigators. Effect of adaptive servo-ventilation on circulating biomarkers in patients with sleep apnoea after myocardial infarction: results of an ancillary analysis of the randomised TEAM-ASV I trial. Sleep Med. 2025 Sep;133:106620. doi: 10.1016/j.sleep.2025.106620. Epub 2025 May 31. PMID 40479758
- [Derived] Summerer V, Arzt M, Fox H, Oldenburg O, Zeman F, Debl K, Buchner S, Stadler S. Occurrence of Coronary Collaterals in Acute Myocardial Infarction and Sleep Apnea. J Am Heart Assoc. 2021 Aug 3;10(15):e020340. doi: 10.1161/JAHA.120.020340. Epub 2021 Jul 30. PMID 34325518
- [Derived] Fox H, Hetzenecker A, Stadler S, Oldenburg O, Hamer OW, Zeman F, Bruch L, Seidel M, Buchner S, Arzt M; TEAM-ASV I Investigators. Rationale and design of the randomised Treatment of sleep apnoea Early After Myocardial infarction with Adaptive Servo-Ventilation trial (TEAM-ASV I). Trials. 2020 Jan 31;21(1):129. doi: 10.1186/s13063-020-4091-z. PMID 32005277